CLINICAL TRIAL: NCT02155270
Title: Impact of a Corneal Pre-cut on Wound Architecture and Astigmatism in Cataract Surgery - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prof.Dr.MBA, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Precut
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Cataract
Keywords: Cataract; Incision; Precut; Corneal; OCT; Intraoperative OCT; Imaging; Astigmatism; Clear corneal incision
MeSH Terms: conditions — Cataract; Surgical Wound; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precut (Active Comparator): A corneal precut of 600µm will be performed.
  Interventions: Procedure: Corneal precut 600µm
- Stab incision (Active Comparator): A stab incision without corneal precut will be performed.
  Interventions: Procedure: Corneal stabincision

INTERVENTIONS:
Procedure: Corneal precut 600µm
  Arms: Precut
Procedure: Corneal stabincision
  Arms: Stab incision

SUMMARY:
We would like to evaluate the use of a 600μm pre-cut regarding wound architecture and surgically induced astigmatism as compared to a stab-incision (a corneal incision without a pre-cut). A dedicated wound architecture score will be used to evaluate wound configuration.

Postoperatively, OCT scans will be obtained, corneal curvature will be measured and subjective and objective refraction will be performed in order to measure the surgically-induced astigmatism.

DETAILED DESCRIPTION:
Corneal wound architecture in cataract surgery has recently been assessed1-4 using optical coherence tomography. However, none of these studies observed the effect of the wound architecture on postoperative astigmatism. In a previous study performed at our center, cataract surgery using a 1.8 mm micro incision (MICS) was compared to a 2.5 mm standard incision (SICS) regarding wound architecture and surgically induced astigmatism. Wound size and wound architecture were assessed using a Time-Domain OCT intraand postoperatively. After implantation of the IOL the incisions were shown to be larger than planned.

This effect was shown to be more pronounced in the small incision group. Both epithelial and endothelial wound gaping at the end of surgery occurred more often in the MICS group. Furthermore, this study showed no effect of a 300 μm pre-cut on postoperative wound architecture and surgically induced astigmatism. Based on these findings we would like to perform another study using a high-resolution Spectral-Domain OCT, which allows for a three-dimensional depiction of wound architecture and a better understanding of the dynamic changes in wound structure during surgery. Furthermore a new high resolution OCT device will be available outside the operating theatre for postoperative measurements. Both devices are CE certified, will be used according to their indication and allow noncontact and therefore pain free measurements. As no significant impact of a 300μm pre-cut on wound architecture and astigmatism was shown in the predecessor study, we would like to evaluate the use of a 600μm pre-cut regarding wound architecture and surgically induced astigmatism as compared to a stab-incision (a corneal incision without a pre-cut). A dedicated wound architecture score will be used to evaluate wound configuration.

Postoperatively, OCT scans will be obtained, corneal curvature will be measured and subjective and objective refraction will be performed in order to measure the surgically-induced astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Age 21 and older
* written informed consent prior to recruitment

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Any ophthalmic abnormality that could compromise the measurements

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Correlation between a wound architecture score and the post-operative astigmatism for the "pre-cut" group and the "stab-incision" group | 1 month

SECONDARY OUTCOMES:
Morphological changes over time | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, MBA, Principal Investigator — VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital Vienna, Vienna, Austria 1140
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Austria

REFERENCES:
- [Derived] Doeller B, Hirnschall N, Fichtenbaum M, Nguyen PM, Varsits R, Findl O. A Randomized Study of the Impact of a Corneal Pre-Cut During Cataract Surgery on Wound Architecture and Corneal Astigmatism. Ophthalmol Ther. 2021 Jun;10(2):313-320. doi: 10.1007/s40123-021-00339-0. Epub 2021 Mar 11. PMID 33709325